CLINICAL TRIAL: NCT05570305
Title: A Study to Assess the Effects of the Endothelin Receptor Antagonist Zibotentan and the SGLT2 Inhibitor Dapagliflozin in Patients With Type 2 Diabetes and Elevated Albuminuria: a Randomized Double Blind Cross-Over Trial
Brief Title: Zibotentan and Dapagliflozin in Patients With Type 2 Diabetes and Elevated Albuminuria
Acronym: ZODIAC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 202100178; 2021-001324-18 (EudraCT Number)
Record Dates: First submitted 2022-10-05; First posted 2022-10-06 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Chronic Kidney Diseases
Keywords: Diabetic Nephropathies; Albuminuria; Chronic kidney disease; Endothelin receptor antagonists; Sodium Glucose Co Transporter 2 inhibitors
MeSH Terms: conditions — Renal Insufficiency, Chronic; Diabetic Nephropathies; Albuminuria | interventions — ZD4054; dapagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The first and second treatment period are double-blind, whereas the final and third treatment period (dapagliflozin and zibotentan) is open-label.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment order 1 (Experimental): Subjects will start with 4 weeks of placebo in treatment period one, then 4 weeks of zibotentan during treatment period two. The order of the first two treatment periods is random which means that patients can start with either placebo or zibotentan. Then in treatment period three, patients are randomized to either either placebo or dapagliflozin for 2 weeks followed immediately by 4 weeks of both zibotentan and dapagliflozin. Between treatment periods there is a 4-week wash-out.
  Interventions: Drug: Zibotentan; Drug: Dapagliflozin; Drug: Placebo; Drug: Dapagliflozin and Zibotentan
- Treatment order 2 (Experimental): Subjects will start with 4 weeks of dapagliflozine in treatment period one, then 4 weeks of zibotentan during treatment period two. The order of the first two treatment periods is random which means that patients can start with either dapagliflozine or zibotentan. Then in treatment period three, patients are randomized to either either placebo or dapagliflozin for 2 weeks followed immediately by 4 weeks of both zibotentan and dapagliflozin. Between treatment periods there is a 4-week wash-out.
  Interventions: Drug: Zibotentan; Drug: Dapagliflozin; Drug: Placebo; Drug: Dapagliflozin and Zibotentan

INTERVENTIONS:
Drug: Zibotentan — Zibotentan 1.5 mg once per day as a hard capsule.
Drug: Dapagliflozin — Dapagliflozin 10 mg once per day as a tablet.
Drug: Placebo — Matching placebo.
Drug: Dapagliflozin and Zibotentan — Dapagliflozin 10 mg once per day as a tablet in combination with zibotentan 1.5 mg once per day as a hard capsule.

SUMMARY:
The aim of this study is to test the hypothesis that the effects on albuminuria of combination treatment with the endothelin receptor antagonist zibotentan and SGLT2i dapagliflozin are complimentary and additive while the fluid retaining effects of zibotentan can be mitigated by dapagliflozin.

DETAILED DESCRIPTION:
A double-blind randomized placebo controlled cross-over study will be conducted in male and female subjects with type 2 diabetes aged between 18 and 75 years, urinary albumin:creatinine ratio (UACR) levels between 100 and 3500 mg/g, and an eGFR ≥ 30 ml/min/1.73m2 will be enrolled. Patients with type 1 diabetes or non-diabetic kidney disease will be excluded.

The study will consist of a screening visit, a 4-week (up to a maximum of 16-weeks) run-in phase for those subjects not on stable ACEi/ARB treatment. Subjects will be randomly assigned to one of two treatment orders. Each treatment order consists of three treatment periods, separed separated by 4-week wash-out period. Treatment period 1 and 2 take four weeks. The third treatment period last 6 weeks.

Participants will be randomized to treatments in addition to receiving background local standard of care (SoC) therapy as follows:

1. Zibotentan 1.5 mg once daily + Dapagliflozin 10 mg once daily.
2. Zibotentan 1.5 mg once daily.
3. Dapagliflozin 10 mg once daily.
4. Placebo once daily.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 and ≤75 years
* Urinary albumin:creatinine ratio > 100 mg/g and ≤ 3500 mg/g in a first morning void urine collection
* eGFR ≥ 30 mL/min/1.73m2
* On a stable dose of an ACEi or ARB for at least 4 weeks prior to randomization
* Willing to sign informed consent

Exclusion Criteria:

* Diagnosis of type 1 diabetes
* Minimal change disease, unstable rapidly progressing renal disease, and/or renal disease requiring significant immunosuppression, autosomal dominant or autosomal recessive polycystic kidney disease
* Hba1c > 12.5%
* Urinary protein excretion > 3500 mg/day
* Heart Failure NYHA Class III or IV
* NT-proBNP > 600 pg/ml
* Hemoglobin <9g/dL
* Acute coronary syndrome event within the preceding 6 months
* Severe peripheral edema according to investigators opinion
* Women of childbearing potential (WOCBP). WOCBP is defined as women who have experienced menarche and who have not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or who are not post-menopausal
* Pregnancy or breastfeeding
* Indication for immunosuppressants according to Investigator's opinion
* Active malignancy aside from treated squamous cell or basal cell carcinoma of the skin within the last 5 years.
* Use of the co-interventional treatments (outlined in section 5.2) within 6 weeks of screening.
* Any medication, surgical or medical condition which might significantly alter the absorption, distribution, metabolism, or excretion of medications including, but not limited to any of the following:

  * History of active inflammatory bowel disease within the last six months;
  * Major gastrointestinal tract surgery such as gastrectomy, gastroenterostomy, or bowel resection;
  * Gastro-intestinal ulcers and/or gastrointestinal or rectal bleeding within last six months;
  * Pancreatic injury or pancreatitis within the last six months;
  * Evidence of hepatic disease as determined by any one of the following: ALT or AST values exceeding 3x ULN at the screening visit, a history of hepatic encephalopathy, a history of esophageal varices, or a history of portocaval shunt;
  * Evidence of urinary obstruction or difficulty in voiding at screening
* Severe hepatic impairment
* History of epilepsy syndrome
* History of severe hypersensitivity or contraindications to dapagliflozin
* History of hypersensitivity or contraindications to iodinated contrast media
* Subject who, in the assessment of the investigator, may be at risk for dehydration or volume depletion that may affect the interpretation of efficacy or safety data
* Participation in any clinical investigation within 3 months prior to initial dosing.
* Donation or loss of 400 ml or more of blood within 8 weeks prior to initial dosing.
* History of drug or alcohol abuse within the 12 months prior to dosing, or according to investigator's assessment.
* History of noncompliance to medical regimens or unwillingness to comply with the study protocol.
* Any surgical or medical condition, which in the opinion of the investigator, may place the patient at higher risk from his/her participation in the study, or is likely to prevent the patient from complying with the requirements of the study or completing the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2022-10-06 (Actual); Primary Completion 2025-03-05 (Actual); Study Completion 2025-03-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline in albuminuria after 4 weeks combined zibotentan and dapagliflozin treatment versus four weeks treatment with zibotentan alone. | The albuminuria will be measured before start of medication intake and after the last intake of medication for each treatment period. This concerns a 4 week time frame.
  The change in albuminuria as expressed the percentage change of the log-transformed albumin:creatinine ratio in mg/gram. The log-transformation is because of the skewed distribution.

SECONDARY OUTCOMES:
Change in Extracellular Fluid | 4 weeks
  Extracellular Fluid measured by bioimpedance spectroscopy
Change in bodyweight | 4 weeks
  Change in kilograms
Change in NT-proBNP | 4 weeks
  N-terminal B-type natriuretic peptide (NT-proBNP)
Change in BNP | 4 weeks
  B-type natriuretic peptide (BNP)
Change in Glomerular Filtration Rate (GFR) | 4 weeks
  Glomerular Filtration Rate (GFR) using iohexol clearance techniques.
Change in Extracellular volume (ECV) | 4 weeks
  Extracellular volume (ECV) using iohexol clearance techniques.
Change in hematocrit | 4 weeks
  The percentage of red blood cells in blood
Change in systolic and diastolic blood pressure | 4 weeks
  Change in blood pressure as measure in mmHg

OTHER OUTCOMES:
Change in renin-angiotensin-aldosterone system (RAAS) markers | 4 weeks
  Change in RAAS markers in plasma and urine
Change in copeptin | 4 weeks
  Change in copeptin as a surrogate of vasopressin

CONTACTS AND LOCATIONS:
Overall Officials: Hiddo J Lambers Heerspink, PhD, PharmD, Principal Investigator — University Medical Center Groningen
Locations (7):
- Anschutz Medical Campus, Aurora, Colorado, United States
- Canada (2):
  - Toronto General Hospital, Toronto, Ontario
  - Montreal Clinical Research Institute, Montreal, Quebec
- Steno Diabetes Center, Copenhagen, Gentoft, Denmark
- Netherlands (2):
  - Amsterdam Universitair Academisch Centrum, Amsterdam, North Holland
  - University Medical Center Groningen, Groningen
- Center for Cardiovascular Science, Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: New insights from SONAR indicate adding sodium glucose co-transporter 2 inhibitors to an endothelin receptor antagonist mitigates fluid retention and enhances albuminuria reduction — https://doi.org/10.1016/j.kint.2020.09.026